CLINICAL TRIAL: NCT03820375
Title: Registry Study for the Observation of Patients With ESUS/Cryptogenic Stroke (ESUS = Embolic Stroke of Undetermined Source)
Brief Title: Registry Study for the Observation of Patients With ESUS/Cryptogenic Stroke
Acronym: Catch-up-ESUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Lars Kellert, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: 17-685
Record Dates: First submitted 2019-01-14; First posted 2019-01-29 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Embolic Stroke of Undetermined Source
Keywords: Stroke; ESUS; PFO; PFO closure; ICM
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Up to know, there is no clear diagnostic and therapeutic pathway for patients with embolic stroke of undetermined source (ESUS). This prospective registry study, which follows up adult ESUS patients for 36 months, is intended to provide important data for the detection of an individual approach in ESUS patients based on a structured diagnostic and therapeutic pathway.

DETAILED DESCRIPTION:
The open-label, academic, prospective, monocentric, observational registry-study (Catch-up-ESUS registry study) started in 01/2018. All ESUS-patients (≥18 years) treated in our hospital are included and will be followed up for three years. Depending on age (< 60 years or ≥ 60 years), the patients are processed according to a standardized treatment algorithm designed interdisciplinary by neurologists and cardiologists. An insertable cardiac monitor (ICM) is implanted in all of them by default. Patients < 60 years without evidence of atrial fibrillation and co-existing PFO are planned for PFO closure within 6 months after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Embolic stroke of undetermined source or cryptogenic stroke; defined as: non-lacunar brain infarction without proximal arterial stenosis or cardioembolic source or other etiology (e.g. vasculitis, cervical artery dissection)
* ≥18 years
* written consent to participation in the study register by the patient or the legal guardian or authorised representative at the time of inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (≥18 years) treated in our hospital and diagnosed with an ESUS will be collected.
  An extension to additional centres is planned in the course of the project, if good feasibility can be demonstrated.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of stroke | 36 months
  Detection of recurrence of ischemia in CT or MRT imaging due to new clinical symptoms

SECONDARY OUTCOMES:
Atrial fibrillation detection | 36 months
  Through several long-term ECG or ICM
Frequency of other vascular events depending on therapy (e.g. myocardial infarction, vascular death) | 36 months
periprocedural events through PFO closure | 36 months
  questionnaire with yes or no answer possibilities (stroke, systemic embolism, atrial fibrillation, bleeding complications)
Detection of predictors of recurrence of stroke | 36 months
  questionnaire with yes or no answer possibilities about cardiovascular risk factors (congestive heart failure, Hypertension, Diabetes mellitus, vascular disease) and their therapy (medication)
Collection of predictors for the appearance of atrial fibrillation | 36 months
  by laboratory parameters (proBNP), risk stratification of atrial fibrillation in automatic detection, Left atrium size and flow in transthoracic and/or transesophageal echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Lars Kellert, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Ludwig Maximilians University, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feil K, Heinrich J, Kupper C, Muller K, Laub C, von Falkenhausen AS, Becker R, Wollenweber FA, Kaab S, Sinner MF, Kellert L. Catch-up-ESUS - follow-up in embolic stroke of undetermined source (ESUS) in a prospective, open-label, observational study: study protocol and initial baseline data. BMJ Open. 2019 Dec 9;9(12):e031716. doi: 10.1136/bmjopen-2019-031716. PMID 31822542